CLINICAL TRIAL: NCT03244033
Title: Integrating Contextual Factors Into Clinical Decision Support to Reduce Contextual Error and Improve Outcomes in Ambulatory Care
Brief Title: Integrating Contextual Factors Into Clinical Decision Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Loyola University (Other)
Responsible Party: Principal Investigator, Alan Schwartz, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-0555; R01HS025374 (AHRQ)
Record Dates: First submitted 2017-07-31; First posted 2017-08-09 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-04

CONDITIONS: Medical Errors; Decision Support Systems, Clinical; Diagnostic Errors
Keywords: context; contextual error; contextual care; electronic medical record; clinical decision support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contextual Survey + Contextual CDS (Experimental): Contextual factors obtained from patients in the Contextual Survey along with contextual red flags already stored in the EHR will produce a variety of Contextual Clinical Decision Support, both passive and interruptive alerts.
  Interventions: Other: Contextual clinical decision support; Behavioral: Contextual survey
- Contextual Survey Only (Active Comparator): Contextual factors obtained from patients in the Contextual Survey along with contextual red flags already stored in the EHR will not be used for CDS or to produce alerts.
  Interventions: Behavioral: Contextual survey

INTERVENTIONS:
Other: Contextual clinical decision support — Incorporation of contextual data into EHR clinical decision support alerts
  Arms: Contextual Survey + Contextual CDS
Behavioral: Contextual survey — Patients complete a survey asking about red flags that could signal contextual factors relevant to their care

SUMMARY:
Preventing contextual errors requires heightening clinician responsiveness to clues that there are contextual factors during the clinical encounter, in real time. These clues, termed contextual red flags are evident in two sources: the medical record and from patients directly. An effective intervention would prompt clinicians to determine whether there are underlying contextual factors that could be addressed in the care plan, averting contextual error. This desirable process is termed contextual probing.

While clinical decision support (CDS) has been used to provide physicians with timely biomedical information at the point of care to prevent errors and promote appropriate care, this technology also affords an opportunity to draw physician attention to both contextual red flags and contextual factors in order to avert contextual errors. This study assesses the potential of "contextualized CDS" to improve contextualization of care through a randomized controlled intervention trial, with assessment measures of both patient health care outcomes and averted costs associated with overuse and misuse of medical services. The three hypotheses are that CDS:

1. Reduces contextual error: CDS tools that inform clinicians of contextual factors and prompt them to explore contextual red flags should result in a reduction in contextual error.
2. Improve health care outcomes: Contextualized CDS predicts improved health care outcomes defined as a partial or full resolution of the contextual red flag (e.g. elevated HgB A1c) after the index visit.
3. Reduces avoidable health care costs: Contextualized CDS is associated with a reduction in misuse and overuse of inappropriate or unnecessary medical services.

DETAILED DESCRIPTION:
The term patient context refers to the myriad contextual factors in patients' lives that complicate the application of research evidence to patient care. For instance, the inability of a patient to afford a medication for a particular condition is a contextual factor. Contextual factors can be addressed when correctly identified. Substituting a low cost generic for a high cost brand name medication may enable a patient to afford a medication. Addressing contextual factors in a care plan is termed contextualizing care. Conversely, the failure to address a contextual factor when it is feasible to so is a contextual error, because it results in an inappropriate plan of care. In sum, contextual errors are medical errors caused by inattention to patient context. They are common and linked to both diminished health care outcomes and an increase in health care costs related to overuse and misuse of medical services. These findings were determined using a validated method for coding audio recorded data called Content Coding for Contextualization of Care ("4C") collected during the encounters by both real patients, and by unannounced standardized patients (USPs) employing checklists.

Preventing contextual errors requires heightening clinician responsiveness to clues that there are contextual factors during the clinical encounter, in real time. These clues, termed contextual red flags are evident in two sources: the medical record and from patients directly. An effective intervention would prompt clinicians to determine whether there are underlying contextual factors that could be addressed in the care plan, averting contextual error. This desirable process is termed contextual probing.

While clinical decision support (CDS) has been used to provide physicians with timely biomedical information at the point of care to prevent errors and promote appropriate care, this technology also affords an opportunity to draw physician attention to both contextual red flags and contextual factors in order to avert contextual errors. This study assesses the potential of "contextualized CDS" to improve contextualization of care through a randomized controlled intervention trial, with assessment measures of both patient health care outcomes and averted costs associated with overuse and misuse of medical services. The three hypotheses are that CDS:

1. Reduces contextual error: CDS tools that inform clinicians of contextual factors and prompt them to explore contextual red flags should result in a reduction in contextual error.
2. Improve health care outcomes: Contextualized CDS predicts improved health care outcomes defined as a partial or full resolution of the contextual red flag (e.g. elevated HgB A1c) after the index visit.
3. Reduces avoidable health care costs: Contextualized CDS is associated with a reduction in misuse and overuse of inappropriate or unnecessary medical services.

To test the hypotheses, patients who consent to participate will be randomized to usual care or care enhanced with contextualized CDS. Participants will audio record their visits, and the data will be coded using 4C. They will be followed several months after the index visit for assessment of outcomes by blinded assessors using an established tracking method. In addition, USPs presenting with cases containing complicating contextual factors that if overlooked result in overuse and misuse of medical services, will be employed to assess the third hypothesis, and to supplement the data obtained by observing the effects of contextual alerts on the care of real patients for the first hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult patients presenting to outpatient primary care clinics for scheduled appointments who can be contacted in advance of their appointment and the clinicians (physicians or nurse practitioners) seeing those patients at those visits.

Exclusion Criteria:

* • Patients with emergent or unscheduled visits or who do not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saul J Weiner, MD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiner SJ, Schwartz A, Weaver F, Galanter W, Olender S, Kochendorfer K, Binns-Calvey A, Saini R, Iqbal S, Diaz M, Michelfelder A, Varkey A. Effect of Electronic Health Record Clinical Decision Support on Contextualization of Care: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2238231. doi: 10.1001/jamanetworkopen.2022.38231. PMID 36279133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 570 patients were assessed for eligibility to participate across the clinics at the two sites. 118 declined to participate and were not randomized.
Period: Overall Study
Arm/Group | Contextual Survey + Contextual CDS | Contextual Survey Only
Started | 177 | 275
Completed | 177 | 275
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: (As in participant flow diagram)
Groups:
- Total: Total of all reporting groups
Arm/Group | Contextual Survey + Contextual CDS | Contextual Survey Only | Total
Number analyzed (Participants) | 177 | 275 | 452
Age, Customized [Count of Participants; unit: Participants]
  Adult (18 and older) | 177 | 275 | 452
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 182 | 293
  Male | 66 | 93 | 159
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 177 | 275 | 452
Clinic Site [Count of Participants; unit: Participants]
  Site 1 | 118 | 160 | 278
  Site 2 | 59 | 115 | 174

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Contextual Red Flags
Description: Proportion of red flags noted at index visit that have resolved
Time Frame: 6-9 months following index visit
Population: Red flags identified in visits of participants.
Measure: Count of Units; unit: Red flags
Units Other Than Participants: Red flags
Arm/Group | Contextual Survey + Contextual CDS | Contextual Survey Only
Number analyzed (Participants) | 177 | 275
Number analyzed (Red flags) | 362 | 540
Red flags
  Red flag improved/resolved | 116 | 240
  Red flag worsened | 83 | 99
  Red flag unchanged or mixed | 163 | 201
Statistical Analysis 1: Comparison: Contextual Survey + Contextual CDS vs Contextual Survey Only; Logistic mixed effects regression modeling likelihood of red flag improved/resolved (vs. not) during outcome period with fixed effects of intervention, site, and whether contextual factor was incorporated into care plan, and random effects of patient and provider. Red flags may be clustered in patients; patients are clustered in providers; Test type: Superiority; p = .91, Mixed Models Analysis; Adjusted for site (p<.001) and for whether physician contextualized plan (AOR 2.14, p=.001), and random effects of physician and patient; Odds Ratio (OR) = .97, 96% CI 2-sided [.57 to 1.64]

2. Secondary Outcome: Probing of Contextual Red Flags
Description: Proportion of red flags which the examining physician probes
Time Frame: At index visit
Measure: Count of Units; unit: Red flags
Units Other Than Participants: Red flags
Arm/Group | Contextual Survey + Contextual CDS | Contextual Survey Only
Number analyzed (Participants) | 177 | 275
Number analyzed (Red flags) | 362 | 540
Red flags
  Probed | 215 | 271
  Not probed | 147 | 269
Statistical Analysis 1: Comparison: Contextual Survey + Contextual CDS vs Contextual Survey Only; Logistic mixed effects regression modeling likelihood of provider probing red flag (vs. not) during visit with fixed effects of intervention, site, \whether red flag was select on pre-visit questionnaire, and whether audiorecorder was visible to provider, and random effects of patient and provider. Red flags may be clustered in patients; patients are clustered in providers; Test type: Superiority; p = 0.02, Mixed Models Analysis; Adjusted for site, source of red flag, visible/concealed recorder, and random effects of physician and patient; Odds Ratio (OR) = 2.09, 95% CI 2-sided [1.13 to 3.86] — OR>1 indicates greater likelihood in intervention group vs. control

3. Secondary Outcome: Planning for Contextual Factors
Description: Proportion of contextual factors identified during visit that are incorporated into care plan
Time Frame: At index visit
Measure: Count of Units; unit: Contextual factors
Units Other Than Participants: Contextual factors
Arm/Group | Contextual Survey + Contextual CDS | Contextual Survey Only
Number analyzed (Participants) | 177 | 275
Number analyzed (Contextual factors) | 383 | 509
Contextual factors
  Plan contextualized for factor | 221 | 255
  Plan not contextualized for factor | 162 | 254
Statistical Analysis 1: Comparison: Contextual Survey + Contextual CDS vs Contextual Survey Only; Logistic mixed effects regression modeling likelihood of provider incorporating contextual factor into care plan (vs. not) at visit with fixed effects of intervention, site, whether red flag was select on pre-visit questionnaire, whether audiorecorder was visible to provider, whether factor was identified by provider probe, whether factor was revealed by patient, and random effects of patient and provider. Red flags may be clustered in patients; patients are clustered in providers; Test type: Superiority; p = .006, Mixed Models Analysis; Adjusted for site, source of factor, recorder visible/concealed, and random effects of physician and patient; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.32 to 5.41] — OR > 1 indicates greater likelihood in intervention group vs. control

ADVERSE EVENTS:
Time Frame: At index visit for each patient during the study period.
Arm/Group | Contextual Survey + Contextual CDS | Contextual Survey Only
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/275
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/275
Other Adverse Events (participants affected / at risk) | 0/177 | 0/275

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03244033/Prot_SAP_000.pdf